CLINICAL TRIAL: NCT02795832
Title: A Randomised, Double-blind, Placebo Controlled Study to Determine the Safety, Pharmacokinetics and Efficacy of Topical ZPL-5212372 Ointment Administered BID for up to 2 Weeks in Healthy Subjects and Subjects With Atopic Dermatitis.
Brief Title: A Study to Determine the Safety & Efficacy of ZPL-5212372 in Healthy Subjects and in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ziarco Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ziarcopharma
Record Dates: First submitted 2016-06-06; First posted 2016-06-10 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1a (Experimental): ZPL-5212372 1% w/w Ointment BID
  Interventions: Drug: ZPL-5212372 1% w/w Ointment BID
- Cohort 1b (Placebo Comparator): Placebo Ointment BID
  Interventions: Drug: Placebo Ointment BID
- Cohort 2a (Experimental): ZPL-5212372 1% w/w Ointment BID
  Interventions: Drug: ZPL-5212372 1% w/w Ointment BID
- Cohort 2b (Placebo Comparator): Placebo Ointment BID
  Interventions: Drug: Placebo Ointment BID
- Cohort 3a (Experimental): ZPL-5212372 1% w/w OIntment BID
  Interventions: Drug: ZPL-5212372 1% w/w Ointment BID
- Cohort 3b (Placebo Comparator): Placebo Ointment BID
  Interventions: Drug: Placebo Ointment BID

INTERVENTIONS:
Drug: ZPL-5212372 1% w/w Ointment BID
  Arms: Cohort 1a; Cohort 2a; Cohort 3a
Drug: Placebo Ointment BID
  Arms: Cohort 1b; Cohort 2b; Cohort 3b

SUMMARY:
A Randomised, Adaptive Design, Double-Blind (3rd Party Open), Placebo Controlled, Sequential Group Study to Determine the Safety,Tolerability, Pharmacokinetics and Efficacy of Twice Daily Application of a Topical ZPL-5212372 (1.0% w/w) Ointment Administered for up to 2 Weeks in Adult Healthy Volunteers and Patients with Moderate to Severe Atopic Dermatitis

DETAILED DESCRIPTION:
This study was a randomised, adaptive design, double blind (3rd party open), placebo controlled, sequential group study in both healthy volunteers and patients with moderate to severe AD. This study was divided into 3 separate, sequential cohorts:

* Cohort 1 were to assess safety, toleration and pharmacokinetics (PK) with intensive monitoring as in-patients over 7 days of dosing in healthy volunteers.
* Cohort 2 were to assess safety, toleration and PK with intensive monitoring as in-patients over 7 days of dosing in moderate to severe AD patients.
* Cohort 3 were to assess efficacy, safety, toleration and PK as out-patients over 14 days of dosing in moderate to severe AD patients.

Subjects received 1.0% (w/w) ZPL-5212372 or matched placebo ointment topically, twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, aged between 18 and 55 years, inclusive (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).

or

Males and females aged 18-65 years inclusive with physician documented history or diagnosis of atopic dermatitis for at least 6 months prior to screening. AD should be diagnosed by the Eichenfield revised criteria of Hanifin and Rajka.

For Atopic Dermatitis Patients:

Eczema Area and Severity Index (EASI) of ≥9 and <48 at Screening and an EASI of ≥12 and <48 at Day 1.

An Investigator's Global Assessment (IGA) score ≥ 3 at both Screening and Day 1.

Atopic dermatitis affecting between ≥10 to <40% BSA at Screening and ≥10% to <50% BSA on Day 1.

All Subjects:

Evidence of a personally signed and dated informed consent form, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

For Healthy Subjects

* Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Have tattoos covering areas of skin to be dosed with study ointment.
* Subjects who are hirsute in areas of skin to be dosed with study ointment.
* Subjects who have received treatment with an investigational drug within 3 months prior to screening.

For Atopic Dermatitis Patients:

* AD of such severity (EASI >48) that the subject could not comply with the demands of the study and/or the subject is not a suitable candidate for a placebo-controlled study.
* Have concomitant skin disease or infection (e.g. acne, impetigo) or presence of skin comorbidities in the study area to be dosed that may interfere with study assessments.
* Have received phototherapy (e.g. UVA, UVB or PUVA therapy), or systemic therapy (e.g. immunosuppressants [such as cyclosporine, azathioprine, methotrexate], cytostatics) known or suspected to have an effect on AD, within 4 weeks of the start of the study. All other biologics should not have been used within 3 months of the start of study.
* Have received systemic corticosteroids (e.g. oral, intravenous, intraarticular, rectal) within 4 weeks of the start of the study. Subjects on a stable maintenance dose (over the preceding 3 months) of inhaled or intranasal CS may participate.
* Patients treated with oral antihistamines or topical calcineurin inhibitors or topical steroids within 7 days of starting study; intranasal antihistamines for the treatment of allergic rhinitis are acceptable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Parneix, MD, Study Director — Novartis
Locations (3):
- United Kingdom (3):
  - MAC, Blackpool
  - MAC, Leeds
  - MAC, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (ZPL-5212372); Cohort 2 (ZPL-5212372); Cohort 3 (ZPL-5212372): ZPL-5212372 1% w/w Ointment BID
- Cohort 1 - Placebo; Cohort 2b - Placebo; Cohort 3 - Placebo: Placebo Ointment BID
Period: Overall Study
Arm/Group | Cohort 1 (ZPL-5212372) | Cohort 1 - Placebo | Cohort 2 (ZPL-5212372) | Cohort 2b - Placebo | Cohort 3 (ZPL-5212372) | Cohort 3 - Placebo
Started | 8 | 4 | 8 | 3 | 20 | 10
Completed | 8 | 4 | 8 | 3 | 20 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (ZPL-5212372) | Cohort 1 - Placebo | Cohort 2 (ZPL-5212372) | Cohort 2b - Placebo | Cohort 3 (ZPL-5212372) | Cohort 3 - Placebo | Total
Number analyzed (Participants) | 8 | 4 | 8 | 3 | 20 | 10 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (21.0) | 25.8 (22.5) | 22.3 (4.86) | 32.9 (12.77) | 27.6 (8.41) | 29.2 (5.77) | 26.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 3 | 12 | 4 | 24
  Male | 6 | 2 | 7 | 0 | 8 | 6 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in EASI Score in Cohort 3
Description: The EASI is a validated tool used to measure the severity and extent of atopic eczema (Eczema Area and Severity Index). The body is divided into 4 sections of total skin area: head including neck (10%); arms including extremities (20%); trunk (30%) and legs including extremities (40%). Each area is scored and the 4 scores are combined into the final EASI. The severity parameters are measured on a scale of 0 to 3 (from none to severe). For each section, the percentage area of skin involved with eczema is estimated and transformed into an extent grade from 0 to 6, from 0% of involved skin area with eczema to 90-100% of involved skin area with eczema. The sum of all four severity parameters is calculated for each section of skin and then multiplied by the weight of the respective section. This value is then multiplied by the extent score for that body area. The EASI value can range from 0-72, a higher score indicates more severe disease.
Time Frame: Day 1 and Day 14
Population: Full Analysis set
Measure: Mean (Standard Error); unit: percent change from baseline in EASI
Arm/Group | Cohort 3 (ZPL-5212372) | Cohort 3 - Placebo
Number analyzed (Participants) | 20 | 10
percent change from baseline in EASI
  Observed case: number analyzed (Participants) | 20 | 7
  Observed case | -34.24 (6.288) | -34.29 (10.680)
  Multiple imputations | -34.04 (6.445) | -31.03 (11.207)
  Last observation carried forward | -34.04 (7.564) | -15.77 (10.712)
  Worst case imputation | -33.94 (10.794) | 3.66 (15.286)
Statistical Analysis 1: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Observed case; Test type: Superiority — ANCOVA model was fitted with percent change from baseline to Week 2 in EASI score as the dependent variable. Explanatory variables fitted were: treatment group (ZPL-5212372, placebo) and baseline EASI score as a continuous variable; p = 0.5016, ANCOVA — The 1-sided p-value tests if the ZPL-5212372 LS mean is < the placebo LS mean; Mean Difference (Net) = 0.05, 90% CI 2-sided [-21.24 to 21.34], Standard Error of Mean 12.441
Statistical Analysis 2: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Multiple imputations; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4082, ANCOVA — The 1-sided p-value tests if the ZPL-5212372 LS mean is < the placebo LS mean; Mean Difference (Net) = -3.01, 90% CI 2-sided [-24.39 to 18.36], Standard Error of Mean 12.964
Statistical Analysis 3: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Last observation carried forward; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0878, ANCOVA — The 1-sided p-value tests if the ZPL-5212372 LS mean is < the placebo LS mean; Mean Difference (Net) = -18.27, 90% CI 2-sided [-40.65 to 4.11], Standard Error of Mean 13.138
Statistical Analysis 4: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Worst case imputation; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0275, ANCOVA — The 1-sided p-value tests if the ZPL-5212372 LS mean is < the placebo LS mean; Mean Difference (Net) = -37.60, 90% CI 2-sided [-69.53 to -5.66], Standard Error of Mean 18.748

2. Primary Outcome: Percent Change From Baseline in EASI Score Over Time in Cohort 3 - Observed Case
Description: as for outcome 1
Time Frame: Days 1, 5, 8, 10, and 15
Population: Full Analysis set
Measure: Mean (Standard Error); unit: percent change from baseline in EASI
Arm/Group | Cohort 3 (ZPL-5212372) | Cohort 3 - Placebo
Number analyzed (Participants) | 20 | 10
percent change from baseline in EASI
  Day 5 | -16.68 (5.823) | -4.96 (8.247)
  Day 8: number analyzed (Participants) | 20 | 8
  Day 8 | -27.36 (5.284) | -21.41 (8.358)
  Day 10: number analyzed (Participants) | 20 | 8
  Day 10 | -32.50 (5.339) | -26.49 (8.445)
  Day 15: number analyzed (Participants) | 20 | 7
  Day 15 | -34.24 (6.228) | -34.49 (8.445)
Statistical Analysis 1: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Day 5; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1284, ANCOVA — The 1-sided p-value tests if the ZPL-5212372 LS mean is < the placebo LS mean; Mean Difference (Net) = -11.72, 90% CI 2-sided [-28.85 to 5.51]
Statistical Analysis 2: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Day 8; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2765, ANCOVA — The 1-sided p-value tests if the ZPL-5212372 LS mean is < the placebo LS mean; Mean Difference (Net) = -5.95, 90% CI 2-sided [-22.85 to 10.95]
Statistical Analysis 3: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Day 10; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2765, ANCOVA — The 1-sided p-value tests if the ZPL-5212372 LS mean is < the placebo LS mean; Mean Difference (Net) = -6.01, 90% CI 2-sided [-23.08 to 11.06]
Statistical Analysis 4: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Day 15; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5016, ANCOVA; Mean Difference (Net) = 0.05, 90% CI 2-sided [-21.24 to 21.34]

3. Secondary Outcome: Summary of EASI-50 and EASI-75 Responders at Week 2 - Cohort 3
Description: The proportion of subjects who achieved EASI-50 and EASI-75 responses at Week 2 were compared between treatment groups.
  EASI-50 was defined as a ≥50% reduction from baseline in EASI score at Week 2. EASI-75 was defined as a ≥75% reduction from baseline in EASI score at Week 2.
Time Frame: Day 14
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Cohort 3 (ZPL-5212372) | Cohort 3 - Placebo
Number analyzed (Participants) | 20 | 10
participants
  EASI-50 responder | 7 | 3
  EASI-50 Non-responder | 13 | 7
  EASI-75 responder | 3 | 0
  EASI-75 Non-responder | 17 | 10
Statistical Analysis 1: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; EASI 50; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4789, ANCOVA — The 1-sided p-value tests if the ZPL-5212372 LS mean is < placebo LS mean; Odds Ratio (OR) = 1.55, 90% CI 2-sided [0.28 to 10.75]
Statistical Analysis 2: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; EASI-75; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3000, ANCOVA — The 1-sided p-value tests if the ZPL-5212372 LS mean is < placebo LS mean; Odds Ratio (OR) = 2.00, 90% CI 2-sided [0.24 to 999]

4. Secondary Outcome: Percentage of Responders on Investigators Global Assessment in Cohort 3
Description: The following secondary endpoints were assessed for IGA:
  A subject was considered as having IGA success if they achieved a score of 'Clear' or 'Almost clear'; note, as subjects required a score of ≥3 to enter the study they must have had a reduction of ≥2 from baseline to achieve success A subject was considered as having an IGA response if they achieved a score of 'Clear' or 'Almost clear', or a reduction of ≥2 from baseline IGA was summarized for the FAS with counts and percentages by treatment at each visit.
Time Frame: Day 14
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Cohort 3 (ZPL-5212372) | Cohort 3 - Placebo
Number analyzed (Participants) | 20 | 10
Percentage of responders | 5.0 [0.13 to 24.87] | 10.0 [0.25 to 44.50]
Statistical Analysis 1: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Test type: Superiority; p = 0.500, Shapiro-Wilkes test — Results for the ZPL-5212372 and placebo groups are estimated adjusted LS means from the fitted model; The p-value tests if the residuals are normally distributed; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.01 to 19.20]

5. Secondary Outcome: Change From Baseline in NRS for Pruritus at Week 2 - Observed Case in Cohort 3
Description: Numerical Rating Scale (NRS) for Pruritus (worst itch). The Pruritus NRS is an assessment tool that will be used to assess the subject's worst itch as a result of AD in the previous 24 hours.
  They will be asked the following question:
  On a scale of 0 (No Itching) to 10 (Itching as bad as you can imagine), please rate the WORST itching that you felt over the last 24 hours.
Time Frame: Day 1 to day 14
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cohort 3 (ZPL-5212372) | Cohort 3 - Placebo
Number analyzed (Participants) | 20 | 10
score on a scale | -2.46 (0.692) | -2.54 (1.075)
Statistical Analysis 1: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Test type: Superiority; p = 0.5233, Shapiro-Wilkes test; Mean Difference (Net) = 0.07, 90% CI 2-sided [-2.02 to 2.16], Standard Deviation 1.220

6. Secondary Outcome: Summary of Patient Global Impression of Change and Logistic Regression of Patient Global Impression of Change in Cohort 3
Description: Patient Global Impression of Change (PGIC) The PGIC scores were summarised for the FAS with counts and percentages in each treatment group. All data collected were included.
  The PGIC was dichotomized into responders, defined as responses of 'Very Much Improved', 'Much Improved' or 'Minimally improved' and non-responders (all other responses plus missing data).
Time Frame: End of treatment (day 15)
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3 (ZPL-5212372) | Cohort 3 - Placebo
Number analyzed (Participants) | 20 | 10
Participants
  Very much improved | 4 | 1
  Much improved | 5 | 1
  Minimally improved | 7 | 4
  No change | 3 | 1
  Minimally worse | 1 | 1
  Much worse | 0 | 2
  Very much worse | 0 | 0
  Missing | 0 | 0
Statistical Analysis 1: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Test type: Superiority; p = 0.2455, t-test, 1 sided; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.45 to 13.26]

7. Secondary Outcome: Change From Baseline in Body Surface Area at Week 2 - Observed Case in Cohort 3
Description: Body Surface Area (BSA). The percentage BSA affected was summarised at each visit, including change from baseline, by treatment group, using the Full Analysis Set.
Time Frame: Day 1 to day 14
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cohort 3 (ZPL-5212372) | Cohort 3 - Placebo
Number analyzed (Participants) | 20 | 10
score on a scale | -6.26 (2.588) | -3.61 (4.075)
Statistical Analysis 1: Comparison: Cohort 3 (ZPL-5212372) vs Cohort 3 - Placebo; Test type: Superiority; p = 0.2812, Shapiro-Wilkes test — The 1-sided p-value tests if the ZPL-5212372 LS mean is < placebo LS mean; Mean Difference (Net) = -2.66, 90% CI 2-sided [-10.40 to 5.09], Standard Error of Mean 4.521

8. Other Pre Specified Outcome: ZPL-5212372 Cmax for Patients in Cohort 2
Description: PK parameters for patients who had ointment applied over 40% BSA.
Time Frame: Day 1, Day 7
Population: Pharmacokinetic analysis set
Measure: Median (Full Range); unit: pg/mL
Groups:
- Day 1 - Cohort 2 (ZPL-5212372); Day 7 - Cohort 2 (ZPL-5212372): ZPL-5212372 1% w/w Ointment BID
Arm/Group | Day 1 - Cohort 2 (ZPL-5212372) | Day 7 - Cohort 2 (ZPL-5212372)
Number analyzed (Participants) | 1 | 6
pg/mL | 300.6 [300.6 to 300.6] | 135.3 [69.31 to 495.2]

9. Other Pre Specified Outcome: ZPL-5212372 AUCt for Patients in Cohort 2
Description: PK parameters for patients who had ointment applied over 40% BSA.
Time Frame: Day 1, Day 7
Population: Pharmacokinetic analysis set
Measure: Median (Full Range); unit: h*pg/mL
Groups:
- Day17 - Cohort 2 (ZPL-32123721); Day 7 - Cohort 2 (ZPL-32123721): ZPL-5212372 1% w/w Ointment BID
Arm/Group | Day17 - Cohort 2 (ZPL-32123721) | Day 7 - Cohort 2 (ZPL-32123721)
Number analyzed (Participants) | 1 | 6
h*pg/mL | 1301 [1301 to 1301] | 1249 [139.2 to 4789]

10. Other Pre Specified Outcome: ZPL-5212372 Trough Plasma Concentrations in Cohort 3
Description: PK parameters for patients who had ointment applied over 40% BSA.
Time Frame: Day 5, Day 8, Day 10, Day 15
Population: Pharmacokinetic analysis set
Measure: Median (Full Range); unit: pg/mL
Groups:
- Day 5; Day 8; Day 10; Day 15: ZPL-5212372 trough plasma concentrations
Arm/Group | Day 5 | Day 8 | Day 10 | Day 15
Number analyzed (Participants) | 20 | 20 | 19 | 20
pg/mL | 88.985 [0.00 to 644.39] | 114.700 [0.00 to 380.42] | 113.920 [0.00 to 287.07] | 90.825 [0.00 to 456.01]

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 56 days. All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 9 months.
Groups:
- Cohort 1 ZPL-5212372 10% BSA: Cohort 1 ZPL-5212372 10% BSA
- Cohort 1 ZPL-5212372 40% BSA: Cohort 1 ZPL-5212372 40% BSA
- Cohort 1 Placebo 10% BSA: Cohort 1 Placebo 10% BSA
- Cohort 1 Placebo 40% BSA: Cohort 1 Placebo 40% BSA
- Cohort 2 ZPL-5212372 10% BSA: Cohort 2 ZPL-5212372 10% BSA
- Cohort 2 ZPL-5212372 40% BSA: Cohort 2 ZPL-5212372 40% BSA
- Cohort 2 Placebo 10% BSA: Cohort 2 Placebo 10% BSA
- Cohort 2 Placebo 40% BSA: Cohort 2 Placebo 40% BSA
- Cohort 3 ZPL-5212372: Cohort 3 ZPL-5212372
- Cohort 3 Placebo: Cohort 3 Placebo
Arm/Group | Cohort 1 ZPL-5212372 10% BSA | Cohort 1 ZPL-5212372 40% BSA | Cohort 1 Placebo 10% BSA | Cohort 1 Placebo 40% BSA | Cohort 2 ZPL-5212372 10% BSA | Cohort 2 ZPL-5212372 40% BSA | Cohort 2 Placebo 10% BSA | Cohort 2 Placebo 40% BSA | Cohort 3 ZPL-5212372 | Cohort 3 Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6 | 0/1 | 0/3 | 0/2 | 0/6 | 0/1 | 0/2 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6 | 0/1 | 0/3 | 0/2 | 0/6 | 0/1 | 0/2 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 2/2 | 3/6 | 1/1 | 1/3 | 2/2 | 4/6 | 1/1 | 2/2 | 17/20 | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 ZPL-5212372 10% BSA (N=2) | Cohort 1 ZPL-5212372 40% BSA (N=6) | Cohort 1 Placebo 10% BSA (N=1) | Cohort 1 Placebo 40% BSA (N=3) | Cohort 2 ZPL-5212372 10% BSA (N=2) | Cohort 2 ZPL-5212372 40% BSA (N=6) | Cohort 2 Placebo 10% BSA (N=1) | Cohort 2 Placebo 40% BSA (N=2) | Cohort 3 ZPL-5212372 (N=20) | Cohort 3 Placebo (N=10)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
NEUTROPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
APPLICATION SITE PARAESTHESIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CATHETER SITE HAEMATOMA (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
FEELING ABNORMAL (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
PARONYCHIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ACNE (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 6
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
REBOUND ATOPIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SKIN BURNING SENSATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
TOOTH EXTRACTION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT02795832/SAP_000.pdf
  • Study Protocol (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT02795832/Prot_001.pdf